CLINICAL TRIAL: NCT02414308
Title: The Role of Adipose Tissue Stem Cell Injection Through Corpora Cavernosa and Intra Dorsal Penile Artery in Management of Erectile Dysfunction Associated With Peyronie's Disease
Brief Title: Management of Peyronie's Disease With Adipose Tissue Stem Cell
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Man Clinic for Andrology, Male Infertility and Sexual Dysfunction (Other)
Responsible Party: Principal Investigator, Khaled Abdulmoneim Gadalla, Dr, Man Clinic for Andrology, Male Infertility and Sexual Dysfunction
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2014-01-06; First posted 2015-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Erectile Dysfunction; Peyronie' Disease
Keywords: Erectile dysfunction, Peyronie's disease, stem cell
MeSH Terms: conditions — Erectile Dysfunction; Balanitis Xerotica Obliterans; Penile Induration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adipose tissue stem cell injection (Experimental): The stem cell will be harvested by liposuction and injection will be at corpora cavernosa and dorsal penile artery
  Interventions: Drug: Adipose tissue stem cell injection

INTERVENTIONS:
Drug: Adipose tissue stem cell injection — Stem cell will be harvested through adipose tissue by liposuction and isolation occurred Injection will distribute through corpora cavernosa and dorsal penile artery

SUMMARY:
Erectile dysfunction is growing in prevalence all over the world and one of the most existing disease in old age patients There is many lines of treatment concerning the status of patient like psychosexual, medical, and surgical treatment But Pyronie's disease is common now among people especially diabetics, and the role of treatment still controversial in results We can start conservative treatment and then surgical treatment if fail but the outcome still not convinced Many patients refuse to fix penile prosthesis and to make operation like nesbite for probability of shortening of penis We start to use stem cell in patients have erectile dysfunction and Peyronie's disease The injection of stem cell will be at corpora cavernosa and intra dorsal penile artery under Doppler device guidance

DETAILED DESCRIPTION:
Peyronie's disease associated with erectile dysfunction nan be treated by different methods We start to treat such patients with adipose tissue stem cell Harvesting stem cell from adipose tissue and injected into corpora cavernosa and penile artery and we assess quality of erection through patient history and penile duplex and also assess plaque size and other symptoms related to Peyronie's disease

ELIGIBILITY:
Inclusion Criteria:

* erectile dysfunction associated with Peyroni's diseas

Exclusion Criteria:

* nil

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-05 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
sexual function questionnaire | 2-3 months
  Clinical history of patients before and after treatment Penile duplex study

SECONDARY OUTCOMES:
Penile plaque assessment | 2-3 months
  Clinical examination Patient history Penile duplex

CONTACTS AND LOCATIONS:
Overall Officials: Khaled A Gadalla, MD, ABS, Principal Investigator — Man clinic
Locations (2):
- Egypt (2):
  - Man clinic for andrology and male infertility, Cairo, Cairo Governorate
  - Man clinic, Cairo